CLINICAL TRIAL: NCT05752734
Title: Preoperative Dexamethasone Enhances Quality of Recovery After Laparoscopic Bariatric Surgery: A Prospective Observational Study
Brief Title: Preoperative Dexamethasone to Improve Quality of Recovery After Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Yasemin Burcu Ustun, Professor, Ondokuz Mayıs University
Other Study IDs: SLGQR402022
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia; Analgesia; Acute Pain
Keywords: dexamethasone; quality of recovery-40; acute pain scores; morphine consumption
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D: Patients who used/applied dexamethasone before bariatric surgery were included in this group.
  Interventions: Drug: Group D
- Group C: Patients who did not use dexamethasone or steroid-derived drugs were included in this group.
  Interventions: Drug: Group C

INTERVENTIONS:
Drug: Group D — Patients who received 8 mg dexamethasone before bariatric surgery will be included in this group.
  Multimodal analgesia protocol is applied to all patients undergoing bariatric surgery in our clinic. According to this protocol, patients are administered iv tenoxicam 20mg, tramadol 100mg after induction of general anesthesia, and iv morphine (0.05mg/kg/IBW) intraoperatively. Postoperative analgesia: iv paracetamol 1gr every 8 hours and iv pca of 0,4mg/ml morphine (the bolus dose is 1mg, the lock-in time of 15 minutes, the 4-hour limit is adjusted to be 40% of the calculated total dose). In cases where rescue analgesia is required (VAS score ≥3) 0.5 mg/kg tramadol is administered to patients. For postoperative nausea and vomiting prophylaxis, patients are routinely administered ondansetron 4 mg IV 20 minutes before extubation.
  Other Names: dexamethasone group
  Groups: Group D
Drug: Group C — Patients not administered dexamethasone will be included in this group.
  Multimodal analgesia protocol is applied to all patients undergoing bariatric surgery in our clinic. According to this protocol, patients are administered iv tenoxicam 20mg, tramadol 100mg after induction of general anesthesia, and iv morphine (0.05mg/kg/IBW) intraoperatively. Postoperative analgesia: iv paracetamol 1gr every 8 hours and iv pca of 0,4mg/ml morphine (the bolus dose is 1mg, the lock-in time of 15 minutes, the 4-hour limit is adjusted to be 40% of the calculated total dose). In cases where rescue analgesia is required (VAS score ≥3) 0.5 mg/kg tramadol is administered to patients. For postoperative nausea and vomiting prophylaxis, patients are routinely administered ondansetron 4 mg IV 20 minutes before extubation.
  Other Names: control group
  Groups: Group C

SUMMARY:
In the obese patient, adequate pain relief in the postoperative period is an important parameter that affects patient comfort and hospital stay. Increasing patient comfort and recovery quality can be achieved by avoiding undesirable effects such as nausea and vomiting, as well as analgesia. In our study, our aim is to evaluate the effect of dexamethasone added to multimodal analgesia on postoperative patient comfort in the obese patient group with a 40-item scale.

DETAILED DESCRIPTION:
Postoperative pain prolongs hospital stay, delays wound healing, increases infection rates, and increases the incidence of drug side effects due to the use of systemic pain relievers (especially opioids).

Good pain control facilitates respiratory effort, allows the patient to perform respiratory exercises and cough to correct the increased thoracic fat mass and impaired respiratory mechanics due to anesthesia. The patient without pain is mobilized early and discharged early.

Our aim is to evaluate the effect of dexamethasone added to multimodal analgesia on postoperative patient comfort in the obese patient group with a 40-item scale.

Patients will be divided in to two groups (group D and group C):

Group D (Dexamethasone Group):

Patients who used/applied dexamethasone before bariatric surgery were included in this group.

Group C(Control Group):

Patients who did not use dexamethasone or steroid-derived drugs were included in this group.

The patients included in the study were evaluated with the 40-item recovery quality scale (QoR-40) 24 hours after the operation.

İn addition all patients will be administered iv morphine pca (patient controlled analgesia) for the first 24 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Body mass index>30 kg/m2
* The American Society of Anaesthesiologists (ASA) physical status class I, II
* The American Society of Anaesthesiologists (ASA) physical status class III only because of morbid obesity
* Patients who will undergo an elective laparoscopic sleeve gastrectomy (LSG)
* Those who are literate enough to answer the compilation quality score (QoR-40) questionnaire

Exclusion Criteria:

* refusal to participate
* allergy to the study drugs
* chronic kidney disease (creatinine>150 μmol/L)
* mental illness
* liver, respiratory or oncological disease,
* cardiac dysfunction (ejection fraction <40%),
* uncontrolled hypertension,
* preoperative analgesic use,
* chronic pain,
* history of alcohol or drug addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BMI > 30 undergoing elective laparoscopic sleeve gastrectomy (LSG)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Global Quality of Recovery (QoR-40) score in the first 24 hours after surgery | postoperative day 1
  The recovery quality of the patients 24 hours after the operation will be evaluated with the QoR-40 questionnaire. The questionnaire consists of 40 questions that examine five domains of patient recovery using a five point Likert scale: none of the time, some of the time, usually, most of the time, and all of the time. The five domains include physical comfort, pain, physical independence, psychological support, and emotional state.
  As a result of the evaluation, the total score ranges from 40 (worst review quality score) to 200 (best review quality score).
The score for each of the five parameters that make up the QoR-40 questionnaire | postoperative day 1
  It consists of 5 parameters: physical independence score (n = 5), patient support score (n = 7), Physical comfort score (n = 12), emotional state score (n = 9) and pain score (n = 7).

SECONDARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | postoperative day 1
  Morphine consumption in the first 24 hours will be measured. Patients will be able to request opioids via a PCA device when their NRS score ≥3.
The incidences of post-operative nausea and vomiting (PONV) | postoperative day 1
  Post-operative nausea and vomiting (PONV) will be evaluated with a verbal descriptive scale.
  (0 = None at all, 1 = Mild nausea, 2 = Moderate nausea, 3 = Vomiting once, 4 = Vomiting more than once)
Time to first mobilization | Up to 24 hours after surgery.
  The patients first mobilization time after the operation will be recorded.
Time to discharge | Trough hospital stay, an average of 1 week
  The length of hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Burcu Üstün, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuzmayıs University, Samsun, Turkey (Türkiye)